CLINICAL TRIAL: NCT02568020
Title: Mechanisms of Low Protein Diet Supplemented With α-ketoacids on Autophagy and Improving Muscle Wasting in Chronic Kidney Disease: the Role of Autophagy in Muscle Wasting
Brief Title: LPD+α-ketoacids on Autophagy and Improving Muscle Wasting in CKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: YUAN Wei-jie (Other)
Responsible Party: Sponsor-Investigator, YUAN Wei-jie, chief physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Keto-019-IP3
Record Dates: First submitted 2015-09-30; First posted 2015-10-05 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- low-protein diet(LPD) (No Intervention): All patients will be treated with a LPD containing 0.6g protein/kg BW per day and 120-125 kJ/kg BW per day.The patients will be followed-up for one year. The patients will come to the hospital every 4 weeks.
- LPD+KA (Experimental): LPD+KA group will be supplemented with keto-amino acids (Ketosteril®, Fresenius Kabi) at a dosage of one tablet/5kg ideal body weight/day, divided into three doses taken during meals.The patients will be followed-up for one year. The patients will come to the hospital every 4 weeks.
  Interventions: Drug: keto-amino acids

INTERVENTIONS:
Drug: keto-amino acids — Ketosteril®( Fresenius Kabi) will be given at a dosage of one tablet/5kg ideal body weight/day, divided into three doses taken during meals.The patients will be followed-up for one year. The patients will come to the hospital every 4 weeks.
  Other Names: Ketosteril®(Fresenius Kabi)
  Arms: LPD+KA

SUMMARY:
To investigate the effects of different dietary regimens on muscle wasting, insulin/IGF-1 resistance. Further, to explore whether LPD+KA decrease the activation of autophagy associate with insulin/IGF-1 pathway.

DETAILED DESCRIPTION:
1. Dietary assessment: The composition of the diet will be evaluated through questionnaire, and analyzed a computer-based nutritional evaluation with Dieta software.
2. Biochemical data: blood samples will be collected at baseline and every 3 months of routine examination, such as blood routine, biochemistry, HbA1c, Serum IGF-1, CRP, will be measured. Homeostatic model assessment score (HOMA-IR) was recorded.
3. Skeletal muscle assessment: the parameters of skeletal muscle will be assessed before and after dietary intervention for 12 months. Body weight, height, Body mass index, skeletal muscle mass will be measured by Body composition analyzer. Quadriceps strength will be assessed with a seated leg press exercise instrument (Keiser Sport, Fresno, CA, USA) using the five repetition maximum technique. Knee and hip extension power (rate of generating force) will be assessed with a validated leg power instrument (University ofNottingham Medical College, Nottingham, UK). Fatigability will be assessed with the same bilateral leg press exercise used in strength testing.

ELIGIBILITY:
Inclusion Criteria:

* patients agree to participate in this study; age≥18 years and<70years; renal function measured with creatinine clearance<60 and >15 ml/min (three monthly consecutive measurements)；at least 6 months of follow up at our clinic before recruitment and haven't received any diet intervention.

Exclusion Criteria:

* pregnant patients; diabetes; heart or liver failure; a recent myocardial infarction (in the last 12 months); long term immobilization; chronic respiratory failure; cancer; any pharmacological treatment that could modify muscle structure or function such as glucocorticoids or insulin；Contraindications of Ketosteril, such as hypersensitivity to the active substances or to any of the excipients, hypercalcaemia, disturbed amino acid metabolism to the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Body weight assessment | 1 year
  the parameters of skeletal muscle will be assessed before and after dietary intervention for 12 months. Body weight will be measured to calculate Body mass index.
skeletal muscle mass | 1 year
  the parameters of skeletal muscle will be assessed before and after dietary intervention for 12 months. muscle circumference including mid-arm, mid-thigh, and mid-calf circumferences will be assessed.
Quadriceps strength assessment | 1 year
  the parameters of skeletal muscle will be assessed before and after dietary intervention for 12 months. Quadriceps strength will be assessed with a seated leg press exercise instrument (Keiser Sport, Fresno, CA, USA) using the five repetition maximum technique.
Knee and hip extension power assessment | 1 year
  the parameters of skeletal muscle will be assessed before and after dietary intervention for 12 months. Knee and hip extension power (rate of generating force) will be assessed with a validated leg power instrument (University ofNottingham Medical College, Nottingham, UK).
Fatigability assessment | 1 year
  the parameters of skeletal muscle will be assessed before and after dietary intervention for 12 months. Fatigability will be assessed with the same leg power instrument (University ofNottingham Medical College, Nottingham, UK) as used in strength testing.
Height assessment | 1 year
  the parameters of skeletal muscle will be assessed before and after dietary intervention for 12 months. Height will be measured to calculate Body mass index

SECONDARY OUTCOMES:
Dietary assessment | 1 year
  The composition of the diet will be evaluated through questionnaire
computer-based nutritional assessment | 1 year
  analyzed a computer-based nutritional evaluation with Dieta software.
Biochemical data | 1 year
  blood samples will be collected at baseline and every 3 months of routine examination, such as blood routine, biochemistry, HbA1c, Serum IGF-1, CRP, will be measured.
calculate HOMA-IR | 1 year
  Homeostatic model assessment score (HOMA-IR) was recorded.
Safety parameters | 1 year
  Blood routine：including WBC, RBC, Hb, PLT, HCT; Blood biochemistry：including Ca, P, iPTH, albumin, prealbumin, transferrin, creatinine, Bun，CRP Blood fat: cholesterol, triglyceride（VLDL、LDL、HDL）

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Gu L, Wang L, Rong S, Yuan W. Low protein diet supplemented with ketoacids on muscle wasting in chronic kidney disease: A clinical trial. Front Med (Lausanne). 2022 Aug 30;9:949108. doi: 10.3389/fmed.2022.949108. eCollection 2022. PMID 36186800